CLINICAL TRIAL: NCT03130686
Title: A Clinical Evaluation of OMRON Digital Blood Pressure Monitor, HEM-9210T, Blood Pressure Measurement Accuracy Based on Auscultation
Brief Title: A Clinical Evaluation of Omron Digital Blood Pressure Monitor
Status: Completed | Type: Observational
Sponsor: Omron Healthcare Co., Ltd. (Industry)
Collaborators: Biwako Chuo Hospital Japan (Unknown); Shared Care Research and Education Consulting,. Inc. US (Unknown)
Responsible Party: Sponsor
Other Study IDs: HDV-TCD-150311
Record Dates: First submitted 2017-04-17; First posted 2017-04-26 (Actual); Last update posted 2017-04-26 (Actual); Status verified 2017-04

CONDITIONS: Blood Pressure

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

INTERVENTIONS:
Device: OMRON blood pressure monitor HEM-9210T — To measure systolic blood pressure, diastolic blood pressure and pulse rate in patients.

SUMMARY:
The purpose of this study is to measure the blood pressure level of the patients, using a cuff ranged 17 - 50 cm.

ELIGIBILITY:
Inclusion Criteria:

* Upper arm circumference: 17-50cm

Exclusion Criteria:

* Patients who has arrhythmia.
* When body motion is observed during measurement.
* Korotkoff sound is poor quality.
* Patient's arm circumference is outside cuff range.
* Patient's auscultatory systolic blood pressure readings differ by more than 12mmHg. and patient's diastolic blood pressure readings differ by more than 8mmHg.
* Patients stated they did not wish to continue with the study and it is stopped before completion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Resident of a community
Sampling Method: Non-Probability Sample
Enrollment: 92 (Actual)
Dates: Start 2015-12-21 (Actual); Primary Completion 2016-02-18 (Actual); Study Completion 2016-03-31 (Actual)

PRIMARY OUTCOMES:
Verify the accuracy of measure functions of device | 30 days
  The aims of this study was to assess the accuracy of the Omron blood pressure monitor according to the ANSI/AAMI/ISO81060-2:2013. And it is analyzed and evaluated at least 85 patients based on the AAMI/ANSI/ISO81060-2:2013.

CONTACTS AND LOCATIONS:
Locations (1):
- OMRON HEALTHCARE CO., Ltd., Mukō, Japan

IPD SHARING:
Plan to Share IPD: No
No plan to share the data.